CLINICAL TRIAL: NCT04456205
Title: The Clinical Effect of Inhaled Corticosteroid Withdrawal in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Inhaled Corticosteroid Withdrawal in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201908041RIND
Record Dates: First submitted 2020-06-10; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: COPD; Inhaled Corticosteroid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dual Therapy: Dual Therapy (long-acting muscarinic antagonist [LAMA] + long-acting beta-agonist [LABA])
- Triple Therapy: Triple Therapy (inhaled corticosteroid [ICS]/ long-acting beta-agonist [LABA] + long-acting muscarinic antagonist [LAMA])

SUMMARY:
According to the WISDOM study, withdraw of inhaled steroids has no effect on the acute exacerbation of chronic obstructive pulmonary disease (COPD), but the lung function of patients with COPD is significantly reclined. In the subgroup analysis of this study, patients with COPD were found to have continued to use inhaled steroids in patients with eosinophilic leukocytes greater than 400 cells/ul or whom has more than two episodes of exacerbation per year. However, in SUNSET study, it was pointed out that withdraw of inhaled steroids had no effect on lung function in patients with COPD, but it was also found that in patients with COPD, eosinophilic leukocytes in the blood were greater than 300 cells/ul, have a better therapeutic response in steroid inhalation. In addition, some studies have shown that in patients with COPD, a decline in lung function after discontinuation of inhaled steroids can make the patient's clinical symptoms worse and increase the risk of acute exacerbations. However, in other comprehensive analytical studies, there are different outcomes. There is no statistically significant difference in the risk of acute exacerbation in patients with COPD after discontinuation of inhaled steroids.

In past studies, it was noted that inhaled steroids cause an increased risk of pneumonia in patients with COPD. However, in these studies, the diagnosis of pneumonia was only from the clinician's suspicion without clear symptom assessment, laboratory examination, microbiological evidence or imaging assessment. Therefore, further research is needed to assess whether patients are suitable for the reduction of inhaled steroids and the impact of COPD in clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed patients with COPD (at least one lung function test post bronchodilator FEV1/FVC <70% before the start of the study)
* Age ≥ 40 years old
* No acute attack record within half a year
* Triple therapy (dual long-acting inhaled bronchodilator and inhaled steroid) is stable for more than six months.
* Eosinophil count in blood <300 cells/ul
* Clinical symptom assessment CAT score <20

Exclusion Criteria:

* Suspected or diagnosed with asthma
* Age <40 years
* Within half a year, there is a record of moderate to severe acute attacks
* Eosinophil count in blood ≥300 cells/ul
* Clinical symptom assessment CAT score ≥20

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Conformed COPD patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test (FEV1) | 6 months
  Spirometry test with forced expiratory volume in one second (FEV1)
Pulmonary Function Test (FVC) | 6 months
  Spirometry test with forced vital capacity (FVC)
Pulmonary Function Test (FEV1/FVC) | 6 months
  Spirometry test with FEV1/FVC ratio
Frequency of Acute Exacerbation | 6 months
  Sudden worsening of COPD symptoms with out-patient clinic and emergency department visit or hospitalization

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) score | 6 months
  COPD Assessment Test (CAT) score ( a patient-completed questionnaire assessing all aspects of the impact of COPD, including cough, sputum, breathlessness, chest tightness, confidence, activity, sleep and energy levels) provides a score of 0-40 to indicate the impact of COPD.
Modified Medical Research Council (mMRC) Dyspnea Scale | 6 months
  Modified Medical Research Council (mMRC) Dyspnea Scale is consisting of just five items containing statements about the impact of breathlessness on the individual and leading to a grade from 1 to 5. (1. Not troubled by breathless except on strenuous exercise; 2. Short of breath when hurrying on a level or when walking up a slight hill; 3. Walks slower than most people on the level, stops after a mile or so, or stops after 15 min walking at own pace; 4. Stops for breath after walking 100 yards, or after a few minutes on level ground; 5. Too breathless to leave the house, or breathless when dressing/undressing).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Yu Chen, Douliu, Yunlin, Taiwan